CLINICAL TRIAL: NCT03259997
Title: Efficacy of Probiotics on Physical Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Probi AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ProFormance135
Record Dates: First submitted 2017-08-17; First posted 2017-08-24 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Physical Performance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic supplement (Active Comparator)
  Interventions: Dietary Supplement: Probiotic supplement
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic supplement — Probiotic supplement
  Arms: Probiotic supplement
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Efficacy of probiotics on physical performance

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 to 40 years, at the time of signing the informed consent form
* Provides signed and dated informed consent form
* Engaged in competitive sports and regularly training
* Non-anemic, iron-deficient
* Willing to comply with all study procedures and be available for the duration of the study

Exclusion Criteria:

* Use of probiotics
* Use of iron supplementation
* Use of ascorbic acid (Vitamin C) supplementation
* Hypersensitivity to any of the ingredients in the investigational product (IP)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2018-05-09 (Actual); Study Completion 2018-05-09 (Actual)

PRIMARY OUTCOMES:
Metabolic response at standardized workloads during ergometer cycling | 4,8 and 12 weeks
  Change from baseline in metabolic response at standardized workloads during ergometer cycling after 4,8 and 12 weeks of supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Michael Svensson, PhD, Principal Investigator — Umeå University
Locations (1):
- Idrottsmedicinska enheten, Umeå universitet, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No